CLINICAL TRIAL: NCT07051707
Title: A Multicenter, Randomized, Study to Evaluate Safety and Efficacy After Treatment With the dNerva Lung Denervation System in Subjects With Chronic Obstructive Pulmonary Disease (COPD) (AIRFLOW-4)
Brief Title: Evaluating the Safety and Efficacy of TLD in Patients With COPD
Acronym: AIRFLOW-4
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nuvaira, Inc. (Industry)
Collaborators: University of Alabama at Birmingham (Other); Temple Health (Unknown); Ohio State University (Other); Honor Health - Clinical Trials (Unknown); Medical College of Wisconsin (Other); University of Pittsburgh Medical Center (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0836
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-07

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: Device: Targeted Lung Denervation (TLD); Optimal Medical Care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into two arms: Targeted Lung Denervation (TLD) therapy plus standard medical care (Treatment) and standard medical care alone (Control). Randomization will be stratified based on investigational site, participation in a pulmonary rehabilitation maintenance program, and baseline single inhaled long acting bronchodilator (LABA-ICS only).
  Participants randomized to Treatment: will undergo TLD treatment with the dNerva Lung Denervation System while continuing the standard medical care that they were on prior to randomization and followed for 2 years or until study closure, whichever is earlier.
  Participants randomized to Control: will continue the standard medical care that they were on prior to randomization, followed for 1 year, then given the option to receive TLD treatment. Whether treated or not, participants will continue follow-up for 1 year or until study closure, whichever is earlier.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Targeted Lung Denervation (TLD) treatment with standard medical care prior to randomization (Experimental): Targeted Lung Denervation (TLD)Therapy is a bronchoscopically guided, minimally invasive procedure using the Nuvaira™ Lung Denervation System while taking regular maintenance medication that minimally includes a long acting bronchodilator with or without a corticosteroid.
  Interventions: Device: Targeted Lung Denervation (TLD); Drug: Standard medical care
- Continuing the standard medical care prior to randomization (Other): Continuing standard of care COPD maintenance medication that minimally includes LABA/ICS, LAMA/LABA or LABA/LAMA/ICS.
  Interventions: Drug: Standard medical care

INTERVENTIONS:
Device: Targeted Lung Denervation (TLD) — Targeted Lung Denervation (TLD)Therapy is a bronchoscopically guided, minimally invasive procedure using the Nuvaira™ Lung Denervation System.
  Other Names: TLD; TLD Therapy
  Arms: Targeted Lung Denervation (TLD) treatment with standard medical care prior to randomization
Drug: Standard medical care — Continuing standard of care COPD maintenance medication that minimally includes LABA/ICS, LAMA/LABA or LABA/LAMA/ICS.
  Other Names: SOC; COPD Maintenance Medications

SUMMARY:
The dNerva Lung Denervation System is one-time treatment intended to improve breathing in Chronic Obstructive Pulmonary Disease (COPD) patients on standard medical care. The purpose of this study is to confirm the safety and efficacy of the Nuvaira Lung Denervation System in the treatment of COPD.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the superiority of treatment with the dNerva Lung Denervation System on top of standard medical care (Treatment arm) compared to standard medical care alone (Control arm) to improve lung function in COPD participants with high RV and low emphysema.

The secondary objective is to compare other efficacy assessments between the Treatment arm and the Control arm, and to confirm the safety profile of lung denervation.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 40 and ≤ 80 years of age at the time of consent?
* Women of childbearing potential must not be pregnant, evidenced by a negative pregnancy test (blood or urine) pre-treatment, or lactating and agree not to become pregnant for the duration of the study?
* Smoking history of at least 10 pack years?
* Not smoking or using any other inhaled substance (e.g. cigarettes, vaping, cannabis, pipes) for a minimum of 2 months prior to consent and agrees to not start for the duration of the study?
* Resting SpO2 ≥ 89% on room air at the time of screening?
* mMRC ≥ 2; CAT score ≥ 10 at the time of screening?
* Diagnosis of moderate to severe COPD as defined by FEV1/FVC < 70% (post-bronchodilator), FEV1 25-<60% predicted, and PaCO2 < 50 (if FEV1 < 30%)? RV ≥ 175% of predicted and RV/TLC > 55% (post-bronchodilator)?
* Participant is on standard medical care, defined as a minimum of therapy with a long-acting bronchodilator, (LABA, LAMA, LABA/ICS or LAMA/LABA) for at least 2 months prior to consent?
* If participant has participated in a formal pulmonary rehabilitation program recently, program completion must have occurred ≥3 months prior to consent; if in a maintenance program, participant agrees to continue their current program through their 12-month follow-up visit; NOTE: Prior participation in a pulmonary rehabilitation program is not required for inclusion in the study.
* Participant is a candidate for bronchoscopy in the opinion of the investigator or per hospital guidelines and is able to discontinue blood thinning medication peri-procedurally.
* Participant is able and agrees to complete all protocol required baseline and follow up tests and assessments including taking certain medications (e.g., azithromycin, prednisolone/prednisone)?

Exclusion Criteria:

* Body Mass Index (BMI) <18 or >32?
* Participant has an implantable electronic device and has not received appropriate medical clearance?
* Uncontrolled diabetes in the opinion of the investigator?
* 4 or more respiratory related hospitalizations within 1 year of consent?
* Malignancy treated with radiation or chemotherapy within 1 year of consent?
* Participant diagnosed with a dominant non-COPD lung disease, or condition affecting the lungs, which is the main driver of the participant's clinical symptoms (e.g., cystic fibrosis, paradoxical vocal cord motion, eosinophilic granulomatosis with polyangiitis (EGPA), allergic bronchopulmonary aspergillosis, interstitial lung disease or active tuberculosis or Asthma) or has a documented medical history of pneumothorax within 1 year of consent?
* Clinically relevant bronchiectasis, defined as > 1/3 cup mucous expectoration daily?
* Pre-existing diagnosis of pulmonary hypertension, clinical evidence of pulmonary hypertension (e.g., cardiovascular function impairment including peripheral edema) and mPAP ≥25 mmHg at rest by right heart catheterization (or estimated right ventricular systolic pressure >50 mmHg by echocardiogram if no previous right heart catheterization)?
* Myocardial infarction within last 6 months, evidence of life-threatening arrhythmias or acute ischemia, pre-existing documented evidence of a LVEF < 40%, stage C or D (ACC/AHA) or Class III or IV (NYHA) congestive heart failure?
* Surgical procedure(s) on the stomach, esophagus or pancreas performed <2 years of consent, or ongoing related symptoms within the past year?
* Symptomatic gastric motility disorder(s) (e.g., gastroparesis) as evidenced by GCSI score ≥18.0, severe uncontrolled GERD (e.g., refractory heartburn, endoscopic esophagitis) or severe dysphagia (e.g., esophageal stricture, achalasia, esophageal spasm)? NOTE: Participants with a hiatal hernia are allowed if Participant meets all other enrollment criteria.
* Any disease or condition that might interfere with completion of a procedure or this study (e.g., structural esophageal disorder, life expectancy <3 years)?
* Prior lung or chest procedure (e.g., BLVR explant procedure, median sternotomy, bullectomy, lobectomy, segmentectomy or other interventional lung or chest procedure) performed ≤1 year of consent? Participants with lung transplant, BLVR valves, LVRS, metal stents within 5cm of the anticipated treatment location; presence of lung volume reduction valves, coils or other lung implants.
* Daily use of >20 mg of prednisone or its equivalent at the time of consent?
* Known contraindication or allergy to medications required for bronchoscopy or general anesthesia (e.g., lidocaine, atropine, propofol, sevoflurane) that cannot be medically controlled?
* Baseline chest CT scan reveals bronchial anatomy cannot be treated with available catheter sizes; presence of whole lung emphysema ≥20% (-950 HU), single lung emphysema >26% (-950 HU), severe bullous disease (>1/3 hemithorax) or discovery of a mass that requires treatment?
* Participant started taking a monoclonal antibody (mAb), or a PDE3/PDE4 inhibitor less than 6 months prior to screening. (Participants on these medications for less than 6 months must wait until 6 months has passed prior to screening.)?
* Participant is currently enrolled in another drug or interventional clinical trial that has not completed follow-up?

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is improvement in FEV1 at 6 months. | 6 months
  FEV1 will be measured through post bronchodilator (Post-BD) force expiratory volume in 1 second (FEV1) test. Change in FEV1 is defined by a comparison between study arms of the mean change in Post-BD FEV1 based on a linear model for change in Post-BD FEV1 from baseline to 6 months follow-up.

SECONDARY OUTCOMES:
Change in Post-BD FEV1 | 12 months
  A comparison between study arms of the mean change in Post-BD FEV1 based on a linear model for change in Post-BD FEV1, adjusted for baseline Post-BD FEV1
Change in Post-BD RV | 12 months
  A comparison between study arms of the mean change in Post-BD RV based on a linear model for change in Post-BD RV, adjusted for baseline Post-BD RV
Transition Dyspnea Index (TDI) | 12 months
  A comparison between study arms of the proportion of participants with a ≥1 point increase in TDI
Change in SGRQ-C | 12 months
  A comparison between study arms of proportion of participants with ≥4 point decrease in SGRQ-C total score from baseline
Annualized rate of Moderate and Severe COPD Exacerbations | 91 days to 12 months post Study day 0.
  A comparison between study arms of annualized rate of exacerbations based on log-rank tests

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Gerard Criner, MD, Principal Investigator — Temple Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication, ending 36 months following article publication.
Access Criteria: Researchers whose proposed use of the data has been approved by a review committee identified for this purpose will have access to the data required to achieve aims in the approved proposal. Proposals should be directed to pjohnson@nuvaira.com. (Link to be provided).